CLINICAL TRIAL: NCT00225537
Title: Evaluation of 4-Methylumbelliferone for Treatment of Chronic Hepatitis B (HBV) and Chronic Hepatitis C (HCV)
Brief Title: 4-Methylumbelliferone as a Treatment for Chronic HBV/HCV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MTmedical Institute of Health (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); BioMonde Preparations Limited (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UTHSCSA 045-900-246
Record Dates: First submitted 2005-06-30; First posted 2005-09-23 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-04

CONDITIONS: Chronic Hepatitis C; Chronic Hepatitis B
Keywords: hcv; hbv; methylumbelliferone; liver; hepatitis; viral; heparvit; hiv; aids
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis B, Chronic; Hepatitis C; Hepatitis B; Hepatitis; Acquired Immunodeficiency Syndrome | interventions — Hymecromone

INTERVENTIONS:
Drug: 4-Methylumbelliferone (Heparvit®)

SUMMARY:
Open-label studies, anecdotal reports, and in vitro scientific research indicate that 4-methylumbelliferone (active ingredient of the dietary supplement Heparvit®) may prevent and reverse the symptoms and complications of chronic infection with hepatitis B virus (HBV)and hepatitis C virus (HCV). This effect has been observed among naïve patients as well as those who are non-responders to interferon, commonly used as first-line therapy for HBV and HCV. In order to scientifically address the efficacy of this 4-methylumbelliferone on chronic viral hepatitis, a randomized, placebo-controlled, blinded study is needed.

It is hypothesized that 4-methylumbelliferone may reduce the impact and aggressiveness of HBV and HCV upon the liver, thereby slowing the progression to potentially life threatening liver diseases such as cancer and cirrhosis. This is a preliminary study designed to determine any indications under controlled conditions that may warrant further detailed clinical studies.

DETAILED DESCRIPTION:
(i). Chronic hepatitis B

Chronicity of HBV following acute infection is strongly age-related; the majority (90%) of infants acquiring HBV perinatally go on to develop chronic infection, while most persons who acquire HBV later in life resolve their infection [ref 1]. Patients with chronic HBV have a 15-25% lifetime risk of liver cirrhosis and hepatic cancer. An estimated 5,000 people die each year from complications of chronic HBV infection (cirrhosis and hepatocellular carcinoma).

Three drugs have been approved by the Food and Drug Administration (FDA) for treatment of chronic HBV: interferon-α (IFN-α), lamivudine, and adefovir dipivoxil. Only one-third of chronic HBV patients develop a sustained response to IFN-α treatment, and adverse effects are common [ref 2]. Use of the newer orally-administered nucleoside analogues (lamivudine or adefovir dipivoxil) typically causes rapid initial clearance of virus and is associated with fewer adverse effects; however, seroconversion rates are low, and long-term therapy with lamivudine (required for sustained responses) frequently results in resistance [ref 2]. Adefovir dipivoxil has, so far, not shown the high rate of resistance observed with lamivudine, but it is expected that resistance will eventually develop [ref 3]. In summary, major problems with currently approved therapy of HBV include expense, toxicity, and development of resistance.

(ii). Chronic hepatitis C

Chronic viral hepatitis due to hepatitis C is an enormous medical problem, affecting approximately 170 million people worldwide (WHO) [ref 4]. In the U.S., an estimated 2.7 million people suffer from chronic HCV, with 10,000-12,000 deaths per year attributable to the disease (ref 5). Chronic HCV infections in the U.S. are usually acquired through injectable drug use, sexual contact, or receipt of contaminated blood products (before antibody screening was initiated in 1990). Most persons exposed to HCV (75%) develop asymptomatic chronic infection. Eventually, 15%-20% will die of cirrhosis and liver cancer without intervention [ref 4].

Only two drugs are licensed for treatment of chronic hepatitis C: IFN-α (standard or pegylated) and ribavirin. Sustained responses to IFN-α monotherapy have occurred in up to 35% of patients; higher responses can be observed with combination treatment (pegylated IFN-α and ribavirin) [ref 6,7]. Responses to combination therapy is closely linked with HCV genotype (types 2 and 3 most responsive). A significant number of patients relapse or do not respond to standard treatment, and retreatment is typically less effective than initial therapy [ref 8].

(iii). 4-methlyumbelliferone

Umbelliferones (7-hydroxycoumarins) [ref 9] are substances present in many species of plants, especially umbelliferae, fabaceae, and oleaceae, which include such common plants as manna ash, sweet woodruff, German chamomile, celery, parsley, and others. In nature, umbelliferones help protect plants from cellular damage, infestation, trauma, and infection. Their 7-hydroxycoumarin derivatives (4-methylumbelliferones) [ref 10] are used in liver therapy, as reagents, plant growth factors, sunscreens, choleretics, and spasmolytics. They are also used as light-protective agents, in the calibration of medical lasers, and in analytical chemistry for the quantitation of nitric acid.

Products containing 4-methylumbelliferone as their active substance have been available in the USA and Europe since 1990, as dietary supplements (under trade names Heparvit®, Heparmed®, DetoxPro®). These products are promoted as supporting liver function and improving detoxification. In many parts of Europe, products containing 4-methylumbelliferone are also available as drugs, and used as spasmolytics and choleretics [ref 11] (improving liver detoxification systems through increased bile production).

7-hydroxycoumarins are also natural metabolites in the body that play important roles in the metabolism of ethanol, chemotherapeutic drugs, acetaminophen, anabolic steroids, and other hepatotoxic drugs [ref 12]. Indeed, measurement of concentrations of 4-methylumbelliferyl glucuronide (a metabolic product of 4-methylumbelliferone) is a common assay for determining the level of toxicity of liver-toxic drugs [ref 13].

The broad potential medical benefits of 4-methylumbelliferone as a hepatoprotectant, anti-inflammatory agent, chemotherapeutic agent, and antiviral substance have been described [ref 13,14]. More recent studies indicate that 4-methylumbelliferone (and other 7-hydroxycoumarin derivatives) may be effective against Helicobacter pylori [ref 15], several types of cancer [ref 15-19], and Alzheimer's disease [ref 20].

ELIGIBILITY:
Inclusion Criteria:

* Serum ALT at least 1.5x the upper limit of normal
* For chronic HBV: Known positive serum HBeAg for at least 6 months; Presence of HBV DNA in serum
* For chronic HCV: Presence of anti-HCV in serum within 6 months of enrollment; Positive serum HCV RNA (enrollment)
* Written informed consent

Exclusion Criteria:

* Treatment (within past 3 months) with interferon, ribavirin, lamivudine, entecavir, or adefovir dipivoxil
* Current treatment with any drug or dietary supplement that could affect serum transaminase values (e.g., milk thistle)
* Pregnancy or inability to practice contraception in patients capable of bearing or fathering children
* Decompensated liver disease (as indicated by total bilirubin >4 mg/dL; albumin <3 g/dL; prolonged (>2 sec over control) prothrombin time; or history of bleeding esophageal varices, ascites or hepatic encephalopathy)
* Active alcohol use, drug abuse, and/or psychiatric problems that, in the investigator's opinion, could interfere with participation in the study
* Hepatitis D infection (for HBV-infected patients)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-09; Study Completion 2007-08

PRIMARY OUTCOMES:
Reduction of virus in blood to undetectable levels;
Normalization of serum ALT and AST.

SECONDARY OUTCOMES:
Reduced viral loads; Improvement of serum ALT and AST;
Improvement in general health status;
Improvement in serum marker of hepatic fibrosis;
Loss of HBeAg/seroconversion to HBeAb (for HBV patients).

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Leach, Prof. M.D., Principal Investigator — University of Texas Health Science Center : Department of Pediatrics; Anastacio M Hoyumpa, Prof. M.D., Principal Investigator — University of Texas Health Science Center : Medicine -Gastroenterolog; Dubravko Pavlin, PhD, Study Director — University of Texas Health Science Center San Antonio
Locations (1):
- University Health Center Downtown "Brady/Green", 527 North Leona,, San Antonio, Texas, United States

REFERENCES:
- [Background] 1: Epidemiology and Prevention of Vaccine-Preventable Diseases, 7th ed, Eds W. Atkinson, C. Wolfe, 2003, Department of Health and Human Services, Centers for Disease Control and Prevention.
- [Background] Asmuth DM, Nguyen HH, Melcher GP, Cohen SH, Pollard RB. Treatments for hepatitis B. Clin Infect Dis. 2004 Nov 1;39(9):1353-62. doi: 10.1086/425010. Epub 2004 Oct 12. PMID 15494913
- [Background] Shaw T, Bowden S, Locarnini S. Chemotherapy for hepatitis B: new treatment options necessitate reappraisal of traditional endpoints. Gastroenterology. 2002 Dec;123(6):2135-40. doi: 10.1053/gast.2002.37288. No abstract available. PMID 12454868
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] NIH Consensus Statement on Management of Hepatitis C: 2002. NIH Consens State Sci Statements. 2002 Jun 10-12;19(3):1-46. PMID 14768714
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Pearlman BL. Hepatitis C treatment update. Am J Med. 2004 Sep 1;117(5):344-52. doi: 10.1016/j.amjmed.2004.03.024. PMID 15336584
- [Background] 9: Penn State College of Medicine. Hershey, PA: 2004. Cited 2004 Dec 29. Faculty Research Expertise Database. Available from: http://fred.hmc.psu.edu/ds/retrieve/fred/meshdescriptor/D014468
- [Background] 10: Penn State College of Medicine. Hershey, PA: 2004. Cited 2004 Dec 29. Faculty Research Expertise Database. Available from: http://fred.hmc.psu.edu/ds/retrieve/fred/meshdescriptor/D006923
- [Background] Abate A, Dimartino V, Spina P, Costa PL, Lombardo C, Santini A, Del Piano M, Alimonti P. Hymecromone in the treatment of motor disorders of the bile ducts: a multicenter, double-blind, placebo-controlled clinical study. Drugs Exp Clin Res. 2001;27(5-6):223-31. PMID 11951580
- [Background] 12: O'Kennedy R, Thornes RD, editors. Coumarins: Biology, Applications and Mode of Action. West Sussex, England: John Wiley & Sons; 1997. ISBN: 0-471-96997-4
- [Background] Muller MJ, Fenk A, Lautz HU, Selberg O, Canzler H, Balks HJ, von zur Muhlen A, Schmidt E, Schmidt FW. Energy expenditure and substrate metabolism in ethanol-induced liver cirrhosis. Am J Physiol. 1991 Mar;260(3 Pt 1):E338-44. doi: 10.1152/ajpendo.1991.260.3.E338. PMID 2003588
- [Background] Fylaktakidou KC, Hadjipavlou-Litina DJ, Litinas KE, Nicolaides DN. Natural and synthetic coumarin derivatives with anti-inflammatory/ antioxidant activities. Curr Pharm Des. 2004;10(30):3813-33. doi: 10.2174/1381612043382710. PMID 15579073
- [Background] Kawase M, Tanaka T, Sohara Y, Tani S, Sakagami H, Hauer H, Chatterjee SS. Structural requirements of hydroxylated coumarins for in vitro anti-Helicobacter pylori activity. In Vivo. 2003 Sep-Oct;17(5):509-12. PMID 14598616
- [Background] Lacy A, O'Kennedy R. Studies on coumarins and coumarin-related compounds to determine their therapeutic role in the treatment of cancer. Curr Pharm Des. 2004;10(30):3797-811. doi: 10.2174/1381612043382693. PMID 15579072
- [Background] Kudo D, Kon A, Yoshihara S, Kakizaki I, Sasaki M, Endo M, Takagaki K. Effect of a hyaluronan synthase suppressor, 4-methylumbelliferone, on B16F-10 melanoma cell adhesion and locomotion. Biochem Biophys Res Commun. 2004 Sep 3;321(4):783-7. doi: 10.1016/j.bbrc.2004.07.041. PMID 15358095
- [Background] Lopez-Gonzalez JS, Prado-Garcia H, Aguilar-Cazares D, Molina-Guarneros JA, Morales-Fuentes J, Mandoki JJ. Apoptosis and cell cycle disturbances induced by coumarin and 7-hydroxycoumarin on human lung carcinoma cell lines. Lung Cancer. 2004 Mar;43(3):275-83. doi: 10.1016/j.lungcan.2003.09.005. PMID 15165085
- [Background] Rilla K, Pasonen-Seppanen S, Rieppo J, Tammi M, Tammi R. The hyaluronan synthesis inhibitor 4-methylumbelliferone prevents keratinocyte activation and epidermal hyperproliferation induced by epidermal growth factor. J Invest Dermatol. 2004 Oct;123(4):708-14. doi: 10.1111/j.0022-202X.2004.23409.x. PMID 15373776
- [Background] 20: Sun S, Kong LY, Zhang HQ, He SA, Niwa M. The asymmetric synthesis of linear dihydropyrano-coumarins for Alzheimer's disease. Heterocycles 2004;63:271-82.
- [Derived] Salman L, Martinez L, Faddoul G, Manning C, Ali K, Salman M, Vazquez-Padron R. Hyaluronan Inhibition as a Therapeutic Target for Diabetic Kidney Disease: What Is Next? Kidney360. 2023 Jun 1;4(6):e851-e860. doi: 10.34067/KID.0000000000000126. Epub 2023 Apr 14. PMID 37055910